CLINICAL TRIAL: NCT05313139
Title: Surveillance of rVSV-ZEBOV Vaccine-induced Immunity Against Ebola Virus in Previously Vaccinated Health Care Workers < EBOSURV >
Brief Title: Surveillance of Vaccine-induced Immunity Against Ebola in Previously Vaccinated Health Care Workers
Acronym: EBOSURV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: 1521/21
Record Dates: First submitted 2022-03-15; First posted 2022-04-06 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Immune Response

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sampling, 3x10mL Lithium Heparine tubes collected by venipuncture
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Unvaccinated participants: Participants who did received the rVSV-ZEBOV vaccine nor had any prior close contact with EBOV patients nor presenting a travel history to East DRC
- Primary vaccinated participants: Participants who received a first rVSV-ZEBOV vaccine dose as part of the WHO vaccination campaign organized in Goma region (end of 2021), of which vaccination date and brand is known
- Participants vaccinated < 1 year ago (from date of enrollment): Participants who received a rVSV-ZEBOV vaccine dose less than a year prior to inclusion of which vaccination date and brand is known
- Participants vaccinated 1-2 years ago (from date of enrollment): Participants who received a rVSV-ZEBOV vaccine dose between 1-2 years prior to inclusion of which vaccination date and brand is known
- Participants vaccinated 2-3 years ago (from date of enrollment): Participants who received a rVSV-ZEBOV vaccine dose between 2-3 years prior to inclusion of which vaccination date and brand is known
- Participants vaccinated > 3 years ago (from date of enrollment): Participants who received a rVSV-ZEBOV vaccine dose > 3 years prior to inclusion of which vaccination date and brand is known

SUMMARY:
During the previous Ebola virus disease (EVD) outbreaks, the institute National de Recherche Biomédicale (INRB) and other institutional's staff in Democratic Republic of the Congo (DRC) got vaccinated with the rVSV-ZEBOV vaccine. However, the longevity of Ebola virus (EBOV)-specific immune responses after vaccination has not been studied extensively (only 1-2 years) nor comprehensively (only humoral), despite the wide use of this vaccine. With the re-emergence of Ebola in North-Kivu from a previously vaccinated individual, and the new planned vaccination campaign (considering homologous booster doses for previously vaccinated HCW) in light of the new outbreak in Beni, assessing the persistence and quality of vaccine-induced anti-EBOV immune responses is pertinent and timely.

DETAILED DESCRIPTION:
Despite the availability of new effective therapeutics, Ebola Virus Disease (EVD) remains a highly lethal disease, with significant collateral impact on the society. In addition, during the last decades, EVD outbreaks appear to become more and more frequent. The disease, therefore, continues to pose a significant public health concern to many areas in West and Central Africa, most notably in the Democratic Republic of the Congo (DRC), where the majority of outbreaks occur.

Fortunately, safe and effective vaccines are now available and these have become a crucial part of the current outbreak response. Most widely used in the DRC is the rVSV-ZEBOV vaccine (licensed as ErveboTM), which was recently approved for human use by both the US Food and Drug Administration (FDA) and the European Medicines Agency (EMA).

Many questions regarding EVD vaccines in general and rVSV-ZEBOV in particular remain unanswered. Currently, there is no data beyond the 2-year time point for antibody titers and more in depth investigations on IgG subclass restrictions or cellular immunity are lacking. However, previous data from non-human primate (NHP) models collectively indicate that Ebola virus (EBOV)-specific CD4+ T cells play a critical role in generating the protective antibody responses and could therefore play a vital part upon re-challenge or prove a vital predictor of poor immunity generation, durability and vaccine failure. These findings argue for an integrated and comprehensive assessment of both durable circulating nAb as well as memory CD4 T cell responses and B cell compartments to fully assess the quality of the long-lived recall responses after a single dose rVSV-ZEBOV vaccination. In addition, there are no post marketing studies that have assessed long-lived immunity outside of a clinical trial environment in routine vaccination campaigns.

Recent events have showed that acquiring such data is of the utmost importance. During the 10th EVD outbreak in DRC in North-Kivu, a person, previously vaccinated with rVSV-ZEBOV, still developed the disease and even relapsed several months later (9). These unresolved questions on the persistence of anti-EBOV immune responses are therefore highly relevant.

Due to concerns on the durability of the immune response after vaccination with rVSV-ZEBOV, a booster dose might be necessary to adequately protect front line health care workers. In this context, the INRB Goma performed a small pilot survey among their personnel, during which they found low binding antibody titers in their previously vaccinated staff (unpublished results). As in October 2021 a new EVD outbreak in North-Kivu was declared, the INRB Goma, in consultation with WHO, decided to, therefore, revaccinate some of their staff that are part of the outbreak response. This would be the first time that the rVSV-ZEBOV vaccine is administered as a booster dose, and documenting the immune response following boostering will be crucial.

The aim of this study is, therefore, to monitor the persistence of the vaccine induced humoral and cellular immune responses following primary vaccination with Ervebo, among recently and previously vaccinated health care staff at INRB Kinshasa and Goma, who received Ervebo as part of the outbreak response.

General objective To comprehensively assess the quality, durability and boostability of the immune response against EBOV glycoprotein antigen in previously and recently rVSV-ZEBOV vaccinated staff

Specific objectives

* Compare EBOV-specific IgG and neutralizing antibodies (nAb) titres at D28 in primary vaccinated staff, and at <1 year, 1-2 years, and 2-3 years and >3 years after primary vaccination in previously vaccinated staff
* Compare the EBOV-specific memory T and B cell responses at D28 in primary vaccinated staff, and at <1 year, 1-2 years, and 2-3 years and >3 years after primary vaccination in previously vaccinated staff
* To characterize the phenotype and quality of the vaccine-induced B and T cell response (isotypes, cell type, polyfunctionality)
* Describe the correlation between humoral and cellular immunity with regard to strength and durability of response after rVSV-ZEBOV vaccination
* In those receiving a booster dose, assess and compare the level of boostability at <1 year, 1-2 years, 2-3 years and >3 years after primary vaccination
* Identify factors influencing the serological and cellular durability and boostability, and the composite immune index expressed as strong, moderate and limited immunity, by vaccination time strata (recently vaccinated, <1 year, 1-2 years, 2-3 years and >3 years)

Exploratory objectives

- Compare vaccine-induced immunity by vaccination time strata (recently vaccinated, <1 year, 1-2 years, and 2-3 years and >3 years, before and after booster dose ) to immunity obtained after natural infection, using a biobanked EVD survivors' cohort

This is a cross-sectional vaccination serosurvey of health care workers (HCWs) from INRB Kinshasa and INRB Goma that were vaccinated with rVSV-ZEBOV, with a short longitudinal follow-up (D0, D7, D28) restricted to recently vaccinated staff to study boostability.

An Ebola outbreak is currently ongoing in Beni. In response to the outbreak and as part of the immunization program, INRB Goma staff that are processing samples from the outbreak area will be offered to be vaccinated against EVD. Recently vaccinated staff, defined as those receiving primary or booster dose, will also be asked for their willingness to participate in the present study, but then with a short and additional longitudinal follow-up.

In our exploratory objective, the vaccine-induced immunity (by vaccination time strata) will be compared to immunity obtained after natural infection. This will depend on whether a solid matched design can be constructed with the the biobanked EVD survivor's cohort from INRB Kinshasa. Only samples from participants that consented to long-term storage and future Ebola-related research will be used.

Recruitment Strategy A list of vaccine recipients is available, including 568 HCWs who received the rVSV-ZEBOV vaccine. All recipients from this list will be contacted by representatives of one of the study sites for their interest in the study and invited to be included in the study. Recruitment will stop once 45 persons per vaccination time strata (<1 year, 1-2 years, and 2-3 years, and >3 years) are reached.

Recently vaccinated staff will be recruited via the current immunization program in place in DRC. All recipients from this list will be contacted by representatives of the study for their interest in the study. Recruitment will stop once 45 persons per group are reached.

Sample Size and Power The study is a cross-sectional vaccination serosurvey across 'time from vaccination' strata, with a longitudinal follow-up restricted to recently vaccinated staff, amongst 245 participants (unvaccinated (n=20), primary vaccinated (n=45), <1 year (n=45), 1-2 years (n=45), 2-3 years (n=45), >3 years (n=45) after primary vaccination).

General overview of study procedures Previously vaccinated health care workers that agree to participate will be scheduled for a single study visit. For recently vaccinated HCWs, 3 study visits will be organized. For logistical reasons, predefined recruitment days will be organized to pool patient visits as much as possible. Depending on their place of residence, the visit will be performed at either the INRB laboratory in Kinshasa or in Goma. During these visits, a questionnaire at D0, will be filled in by the participants. Blood sample of 3 x 10mL Lithium Heparine tubes will be collected. In case of multiple visits, blood samples will be collected at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to give informed consent for participation in the study
* Subject can be contacted by phone, email or physical address
* Subject is aged 18 years or above
* Subject must have a ID card (or other identification document)

For vaccinated group:

- Subject must be receiving the rVSV-ZEBOV vaccine (first or second dose) at time of inclusion OR has received a first rVSV-ZEBOV vaccine dose prior to inclusion of which vaccination date and brand is known

For unvaccinated group (controls):

Subject must NOT have received the rVSV-ZEBOV vaccine nor had any prior close contact with EBOV patients

Exclusion Criteria:

* Subject was previously diagnosed with EVD
* Subject has any contraindication to venipuncture, as determined by clinical judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care workers from Institut National de Recherche Biomédicale (INRB) Kinshasa and Institut National de Recherche Biomédicale (INRB) Goma, who previously or recently received (primary and booster dose), or did not receive (cf. controls) the rVSV-ZEBOV vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
EBOV glycoprotein (GP)-specific T and B cell Spot Forming Units | Day 0
  EBOV glycoprotein (GP)-specific T and B cell Spot Forming Units (SFU) per 10^6 cells determined by Elipot/Fluorospot assay
EBOV glycoprotein (GP)-specific T and B cell Spot Forming Units | Day 7
  EBOV glycoprotein (GP)-specific T and B cell Spot Forming Units (SFU) per 10^6 cells determined by Elipot/Fluorospot assay
EBOV glycoprotein (GP)-specific T and B cell Spot Forming Units | Day 28
  EBOV glycoprotein (GP)-specific T and B cell Spot Forming Units (SFU) per 10^6 cells determined by Elipot/Fluorospot assay

SECONDARY OUTCOMES:
Geometric mean titers (GMT) of GP-specific IgG and neutralizing antibodies (nAb) | Day 0
  Geometric mean titers (GMT) of GP-specific IgG and neutralizing antibodies (nAb)
Geometric mean titers (GMT) of GP-specific IgG and neutralizing antibodies (nAb) | Day 7
  Geometric mean titers (GMT) of GP-specific IgG and neutralizing antibodies (nAb)
Geometric mean titers (GMT) of GP-specific IgG and neutralizing antibodies (nAb) | Day 28
  Geometric mean titers (GMT) of GP-specific IgG and neutralizing antibodies (nAb)
Seroprevalence status based on GP specific antibodies (Ab) | Day 0
  Seroprevalence status based on GP specific antibodies (Ab)
Seroprevalence status based on GP specific antibodies (Ab) | Day 7
  Seroprevalence status based on GP specific antibodies (Ab)
Seroprevalence status based on GP specific antibodies (Ab) | Day 28
  Seroprevalence status based on GP specific antibodies (Ab)
Phenotypic and isotypic classification of GP-responsive T and B cells, respectively | Day 0
  Phenotypic and isotypic classification of GP-responsive T and B cells, respectively
Phenotypic and isotypic classification of GP-responsive T and B cells, respectively | Day 7
  Phenotypic and isotypic classification of GP-responsive T and B cells, respectively
Phenotypic and isotypic classification of GP-responsive T and B cells, respectively | Day 28
  Phenotypic and isotypic classification of GP-responsive T and B cells, respectively
Correlation coefficients between humoral and cellular responses | Day 0
  Correlation coefficients between humoral and cellular responses
Correlation coefficients between humoral and cellular responses | Day 7
  Correlation coefficients between humoral and cellular responses
Correlation coefficients between humoral and cellular responses | Day 28
  Correlation coefficients between humoral and cellular responses
Effect of age, vaccination history, comorbidities and coinfections on serological and cellular titers and on composite immune index, expressed as strong, moderate and limited immunity | Day 0
  Effect of age, vaccination history, comorbidities and coinfections on serological and cellular titers and on composite immune index, expressed as strong, moderate and limited immunity

CONTACTS AND LOCATIONS:
Overall Officials: Mulangu Sabue, Prof, Study Chair — Institut National de Recherche Biomédicale (INRB), Kinshasa; Kavunga Hugo, Prof, Study Chair — Institut National de Recherche Biomédicale (INRB), Goma; Mukadi Daniel, MD, Study Chair — Institut National de Recherche Biomédicale (INRB), Goma
Locations (2):
- Democratic Republic of the Congo (2):
  - Institut National de Recherche Biomédicale (INRB), Goma
  - Institut National de Recherche Biomédicale (INRB), Kinshasa

IPD SHARING:
Plan to Share IPD: Undecided